CLINICAL TRIAL: NCT00113841
Title: Pilot Study of Curcumin (Diferuloylmethane Derivative) With or Without Bioperine in Patients With Multiple Myeloma
Brief Title: Curcumin (Diferuloylmethane Derivative) With or Without Bioperine in Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0436
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Results first posted 2011-10-19 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Diferuloylmethane Derivative; Curcumin; Bioperine
MeSH Terms: conditions — Multiple Myeloma | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcumin (Experimental): Curcumin starting dose 2 grams orally in 2 divided doses (a.m., p.m.).
  Interventions: Drug: Curcumin
- Curcumin + Bioperine (Experimental): Curcumin starting dose 2 grams orally in 2 divided doses (a.m., p.m.) and Bioperine 5 mg orally twice daily.
  Interventions: Drug: Curcumin; Drug: Bioperine

INTERVENTIONS:
Drug: Curcumin — 2 grams (Capsules) orally in 2 divided doses (a.m., p.m.)
Drug: Bioperine — 5 mg (Tablets) orally twice daily
  Arms: Curcumin + Bioperine

SUMMARY:
Primary Objectives:

1. To evaluate clinical tolerance and response to curcumin alone and in combination with Bioperine in patients with multiple myeloma.
2. To compare the pharmacokinetics and pharmacodynamics of curcumin and curcumin + Bioperine and evaluate the effect of Bioperine on the bioavailability of curcumin.
3. To evaluate the biologic effects of curcumin alone and in combination with Bioperine on the expression of NF-kB and related genes in the Multiple Myeloma (MM) cells.

DETAILED DESCRIPTION:
Curcumin, a yellow substance extracted from the plant Curcuma longa, is commonly used as a food additive. It is a natural anti-inflammatory compound and has shown anti-tumor activity in the laboratory. Bioperine is a pepper extract that increases the absorption of nutrient supplements.

In this study, 6 patients at a time will be randomly assigned (as in the toss of a coin) to one of two groups of 3 patients each. One group (Arm A) will receive curcumin alone. The other group (Arm B) will receive curcumin in combination with Bioperine. There is an equal chance of being in either group. While on study you may receive standard supportive care as appropriate.

Both of the study agents will be taken by mouth two times a day. Each group will have five dose levels of curcumin, starting with the lowest dose. After 6 patients have been enrolled in the first level (3 in each arm), the next group will be treated at a new dose level. You will always receive the same dose during your treatment, which will continue for at least 12 weeks unless there is evidence that the disease has gotten worse or intolerable side effects occur. You may receive treatment up to one year depending on your response to treatment.

You may be treated as outpatient and may receive your treatment at home. You will be asked to return to M. D. Anderson every 4 weeks for evaluation and physical exam.

This is an investigational study. A total of up to 30 evaluable patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who have been previously untreated, are asymptomatic and without serious or imminent complications; or have relapsed or failed treatment with conventional therapy.
* Adequate hematologic, renal, and hepatic functions.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.

Exclusion Criteria:

* Previously untreated patients with high tumor mass; symptomatic or impending fractures.
* Patients with significant cardiac disease.
* Patients with comorbid condition which renders patients at high risk of treatment complications.
* History of significant neurological or psychiatric disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — MDAnderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 11/2004 to 1/2008. All participants were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of 42 patients enrolled, 9 were excluded from the trial prior to group assignment because of screen failure.
Groups:
- Curcumin: Curcumin starting dose 2 grams orally in two divided doses (a.m., p.m.)
Period: Overall Study
Arm/Group | Curcumin | Curcumin + Bioperine
Started | 16 | 17
Completed | 15 | 15
Not Completed | 1 | 2
Not completed — Disease progression | 0 | 2
Not completed — Non-compliant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Curcumin + Bioperine | Total
Number analyzed (Participants) | 16 | 17 | 33
Age Continuous [Median (Full Range); unit: years] | 59 [46 to 78] | 62 [41 to 78] | 59 [41 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of NF-kB Protein Expression in Peripheral Blood Mononuclear Cells From Baseline Through 4 Weeks of Treatment
Description: Percent change of NF-kB =[(expression at 4 weeks- expression at baseline)/expression at baseline]*100%. Bone marrow aspirate/biopsy for expression of NF-kB and related genes/proteins markers at baseline and after 4 weeks.
Time Frame: Baseline through 4 weeks of treatment
Population: All participants in the two arms (Curcumin versus Curcumin plus Bioperine) who received at least 4 weeks of treatment were eligible for outcome evaluation.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Curcumin | Curcumin + Bioperine
Number analyzed (Participants) | 15 | 15
Percent reduction | 21 (37) | 37 (25)
Statistical Analysis 1: Comparison: Curcumin vs Curcumin + Bioperine; Test type: Superiority or Other; p = 0.16, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 years and 2 months
Arm/Group | Curcumin | Curcumin + Bioperine
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 9/16 | 9/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Curcumin (N=16) | Curcumin + Bioperine (N=17)
Appetite decreased (Gastrointestinal disorders) | 0 | 1
Burning in the eyes (Eye disorders) | 0 | 1
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0
Redness of eyes (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 1 | 0
Feeling of fullness with capsules (Gastrointestinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Flushing (General disorders) | 2 | 0
Headache (General disorders) | 2 | 4
Indigestion (Gastrointestinal disorders) | 1 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Queasy feeling (Gastrointestinal disorders) | 1 | 0
Yellow discoloration of finger tips (General disorders) | 2 | 0
Yellow discoloration of sweat (General disorders) | 1 | 0
Yellow discoloration of urine (General disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No